CLINICAL TRIAL: NCT00416143
Title: Bed Rest for Idiopathic Sudden Sensorineural Hearing Loss
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-06-4065-EC-CTIL
Record Dates: First submitted 2006-12-24; First posted 2006-12-27 (Estimated); Last update posted 2006-12-27 (Estimated); Status verified 2006-12

CONDITIONS: Sudden Loss of Hearing
Keywords: Bed rest for idiopathic sudden sensorineural hearing loss
MeSH Terms: conditions — Hearing Loss, Sudden | interventions — Bed Rest; Fumigant 93

INTERVENTIONS:
Procedure: bed rest
Drug: prednisone - oral corticosteroid 1mg/kg/D for 1 week

SUMMARY:
sudden sensorineural hearing loss:

* idiopathic in most cases
* 5-20/100,000 new cases annually in the U.S
* no establishes pathogenesis
* treated with oral steroids in most cases
* ~50% improvement in hearing levels
* bed rest - acceptable treatment, not well investigated

ELIGIBILITY:
Inclusion Criteria:

* patients with sudden sensorineural hearing loss

Exclusion Criteria:

* age less than 16 years
* contraindication for oral steroid treatment
* prior steroid treatment for hearing loss
* pregnent women

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2006-06; Study Completion 2008-12

PRIMARY OUTCOMES:
hearing improvement

CONTACTS AND LOCATIONS:
Overall Officials: Eldar Carmel, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel